CLINICAL TRIAL: NCT00559143
Title: Better Pacing - Biventricular Pacing as Alternative Method in Patients With Disturbances of AV Conduction and Preserved LV Function
Brief Title: Biventricular Alternative Pacing
Acronym: BETTER
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No patients enrolled for long period of time. No scientific interest any more
Sponsor: Medtronic Hellas Medical Devices ΑEE (Industry)
Responsible Party: George Athanasiou/ Senior Field Clinical Research Specialist, Medtronic Hellas Medical Devices ΑEE
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 1111 Version 1.0- 01/May/2007
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Atrioventricular Block
Keywords: AV conduction disturbances; LV function; Biventricular Pacing; Conductance Catheters
MeSH Terms: conditions — Atrioventricular Block | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): DDD(R)-RV pacing
  Interventions: Other: Biventricular Pacing (DDD(R)- BiV)
- 2 (Experimental): DDD(R)- BIV pacing
  Interventions: Other: Biventricular Pacing (DDD(R)- BiV)

INTERVENTIONS:
Other: Biventricular Pacing (DDD(R)- BiV) — Subjects indicated for DDD(R) pacing due to AV conduction disturbances and preserved LV function will receive biventricular pacing DDD(R)- BiV

SUMMARY:
Aim of present study is to examine the short and long-term results of pacing from right ventricular apex and to compare them with those of biventricular pacing.

DETAILED DESCRIPTION:
In this study all subjects to be studied will have atrioventricular conduction disturbances that require permanent artificial pacing. In all subjects a biventricular pacemaker will be implanted. Moreover the subjects will be randomized in a biventricular or conventional pacing mode and will be observed for a long term period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the age of 18 to 75 years with classic indication for permanent artificial pacing in which it is expected very high percentage of ventricular pacing, (pacing systoles constitute the 80% and more of the total).
* Physiologic or mildly affected systolic function of left ventricle, LVEF> 40%.
* Subject is willing and able to comply with the Clinical Investigational Plan and to remain available for follow-up visits, through study closure.
* Subject (or if allowed by local law/regulations: subject's legally authorised representative) is willing and able to sign and date the study Informed Consent.

Exclusion Criteria:

* Subjects with classic indication for Biventricular Pacing - (European Guidelines 2007).
* Permanent atrial fibrillation.
* Cardiovascular surgery within the last three months prior to enrollment.
* Myocardial infarction within the last three months prior to enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-11 (Estimated); Study Completion 2011-07 (Estimated)

PRIMARY OUTCOMES:
Change in End Diastolic Diameter of Left Ventricle with the two different ways of pacing (DDD(R)-RV & DDD(R)-BiV) | two years

SECONDARY OUTCOMES:
Tolerance in the cardiopulmonary stress test, quality of life, LV function and changes of BNP, TNF, interleukin-6, interleukin-12 and oxidant stress. | two years
Assessment of the operation of Left Ventricle at the different pacing types using conductance catheters in a subgroup of patients that will perform a programmed coronary angiography due to investigation of possible coronary artery disease. | two years

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Simantirakis, MD, Principal Investigator — University Hospital of Crete; Panagiotis Vardas, MD, Cardiology Professor, Study Chair — University Hospital of Crete
Locations (1):
- University Hospital of Crete, Heraklion, Crete, Greece